CLINICAL TRIAL: NCT05860816
Title: Facilitators and Barriers to Implementing Pain Neuroscience Education Programmes for the Treatment of Patients With Chronic Pain in Primary Care Physiotherapy Units: the Physiotherapist's Perspective
Brief Title: Facilitators and Barriers in Neuroscience-based Pain Education Programmes in Primary Care Physiotherapy
Status: Active, not recruiting | Type: Observational
Sponsor: Castilla-León Health Service (Other)
Responsible Party: Principal Investigator, Paula Areso, Physiotherapist, Castilla-León Health Service
Other Study IDs: CEIm 2925
Record Dates: First submitted 2023-05-06; First posted 2023-05-16 (Actual); Last update posted 2025-02-17 (Actual); Status verified 2025-02

CONDITIONS: Chronic Primary Pain; Musculoskeletal Pain; Fibromyalgia
Keywords: Primary Health Care; Chronic Pain; Physical Therapies Modalities; Health Education
MeSH Terms: conditions — Chronic Pain; Musculoskeletal Pain; Fibromyalgia; Health Education | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Primary Care Physiotherapists working in the Spanish public health system: A sample of primary care physiotherapists fill out a survey on their knowledge of chronic pain management and the approach they use to treat patients with chronic pain.
  Interventions: Other: Survey

INTERVENTIONS:
Other: Survey — Survey aimed at finding out the barriers and facilitators that Spanish primary care physiotherapists have to implement pain neuroscience-based education programmes in patients with chronic pain.

SUMMARY:
The new approach in pain neuroscience education (PNE) requires specific training for the physiotherapists in charge of applying it. In recent years, public and private initiatives have offered training in different formats, online courses, face to face courses, congresses, that have facilitated access to this knowledge for many professionals. However, this offer lacks a sufficiently deep approach, so that physiotherapists do not develop the necessary skills to put it into practice, in addition to being an area of knowledge in which the concepts need constant updating given the rapid scientific progress.

As with any paradigm shift, there is resistance to change on the part of some professionals, but the extent to which this has a collective impact on the generalization of these interventions is unknown.

From our point of view, lack of training is only one of the aspects that hinder the implementation of PNE. Working conditions (pressure of care, high physiotherapist/population ratios, limited time available) and organizational conditions (dependence on hospital services, lack of vision of this model by the PC team) could be among the main daily difficulties in implementing it.

The main objective of this study is to detect the barriers and facilitators that primary care physiotherapists have to implement programmes based on the new paradigm of pain neuroscience in the treatment of patients with chronic pain.

DETAILED DESCRIPTION:
Introduction: Chronic pain is a complex clinical entity with a growing impact on population health. In the Global Burden of Disease 2019 study, pain and pain-related diseases were the leading cause of disability worldwide, with musculoskeletal problems being the most prevalent. According to the International Association for the Study of Pain (IASP), pain can be defined as "an unpleasant sensory and emotional experience associated with, or similar to that associated with, actual or potential tissue damage". This definition tries to include the different dimensions of pain, evolving from survival-oriented nociceptive pain to neuropathic or neuroplastic pain, more related to processes of central sensitisation, inhibition of downstream modulators or temporary summation of stimuli.

Due to its multidimensional nature, pain management is complex and requires frequent assessments to adjust the interventions needed to maintain the quality of life of individuals. Current scientific evidence supports the implementation of primary care programmes based on pain neuroscience education and therapeutic exercise for chronic pain management. The rationale for these interventions is based on autonomous management of the disease by the patient, through increased knowledge of the neurophysiology of pain, improved functional capacity and an addressing of the psychosocial factors involved. Primary care physiotherapists have been shown to play a key role in the management of chronic pain at community level through the development of such programmes.

However, the implementation of these programmes is a clinical challenge due to the lack of knowledge of the approach to chronic pain, the need for specialised training or the provision of resources by health systems. The aim of this study is to identify facilitators and barriers from the point of view of primary care physiotherapists to implement chronic pain management through primary care programmes based on education and therapeutic exercise.

Study design: A cross-sectional observational study will be carried out in primary care physiotherapists in the Spanish national health system. The survey to be used will be an adaptation to Spanish of the one developed by Wilson et al. Study participants should meet the following inclusion criteria: a) be a physiotherapist working in a primary care setting; and b) have more than 2 years of experience in this context. Not working in the public sector will be considered an exclusion criterion.

Potential participants will be contacted through the nursing directors of each health area (an administrative division of the Spanish health system). Participation will also be promoted through social networks. Information about this study will be also available at the IV National Conference on Physiotherapy in Primary Care, to be held on May 12 and 13, 2023 in Barcelona (Spain).

Variables: Independent variables will be: 1) current situation of the primary care physiotherapist (working conditions), 2) training in pain neuroscience, 3) barriers to implementing the approach and 4) available resources. Dependent variables will be: 1) clinical approach used in the management of chronic pain; and 2) Interventions used by the primary care physiotherapist in the treatment of people with chronic pain.

Data collection: The survey will be administered through Google Forms. Participants will receive information on the basic aspects of the study and will sign an informed consent form before taking the survey. The sample size was set at 323 participants considering a confidence level of 95%, an standard deviation of .5, and a margin of error of 土5%.

Data analysis: Survey data will be exported into Excel for cleaning, then transferred to SPSS (v26, IBM Corp., New York, USA) for analysis. Descriptive statistics (mean, standard deviation, frequency) will be used to summarise demographic/survey data. Univariate logistic regression will examine associations between the training of physiotherapists, the barriers experienced, their clinical setting and their available resources (independent variables) and their competency/use of an approach based on pain neuroscience education (dependent variables). For continuous outcomes, univariate linear regression will be used. Multivariate regressions will be used if relevant covariates exist (identified via p<0.10 in univariate regression analysis). Where appropriate, content or thematic analysis will ensure transparent synthesis of open-ended question data. Themes will be identified via answer coding line-by-line if applicable. Only responses with ≥80% of the data completed will be included.

ELIGIBILITY:
Inclusion Criteria:

* Primary Care Physiotherapists in the Spanish national health system with more than two years of experience.

Exclusion Criteria:

* Less than two years of experience in Primary Care
* Do not work in the public system

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Study participants must meet the following inclusion criteria: a) be a physiotherapist working in a primary care setting; and b) have more than 2 years of work experience in this clinical setting. Participants who do not work in the public sector will be excluded from the study.
Sampling Method: Non-Probability Sample
Enrollment: 123 (Actual)
Dates: Start 2023-05-12 (Actual); Primary Completion 2023-12-30 (Actual); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Association between the characteristics of physiotherapists and their treatment approach in chronic pain. | From May 2023 to November 2023
  Univariate logistic regression between the training of physiotherapists, the barriers experienced, their clinical setting and their available resources (independent variables) and their competency/use of an approach based on pain neuroscience education (dependent variables)

SECONDARY OUTCOMES:
Sample demographics | From May 2023 to November 2023
  Descriptive statistics (mean, standard deviation, frequency) of age, gender, educational level and work experience.

CONTACTS AND LOCATIONS:
Overall Officials: Goretti Aranburu-Guenaga, PT, Study Chair; Tasha Stanton, MSc, PhD, Study Chair — University of South Australia; Felicity A Braithwaite, PhD, Study Chair — University of South Australia; Monique Wilson, PhD C, Study Chair — University of South Australia; Paula Areso-Bóveda, PT, Principal Investigator — Servicio de salud de Castilla y León (SACYL); Héctor Hernández-Lázaro, PT, Study Chair — University of Valladolid
Locations (1):
- Paula Areso, Burgos, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Mills SEE, Nicolson KP, Smith BH. Chronic pain: a review of its epidemiology and associated factors in population-based studies. Br J Anaesth. 2019 Aug;123(2):e273-e283. doi: 10.1016/j.bja.2019.03.023. Epub 2019 May 10. PMID 31079836
- [Background] Raja SN, Carr DB, Cohen M, Finnerup NB, Flor H, Gibson S, Keefe FJ, Mogil JS, Ringkamp M, Sluka KA, Song XJ, Stevens B, Sullivan MD, Tutelman PR, Ushida T, Vader K. The revised International Association for the Study of Pain definition of pain: concepts, challenges, and compromises. Pain. 2020 Sep 1;161(9):1976-1982. doi: 10.1097/j.pain.0000000000001939. PMID 32694387
- [Background] Cieza A, Causey K, Kamenov K, Hanson SW, Chatterji S, Vos T. Global estimates of the need for rehabilitation based on the Global Burden of Disease study 2019: a systematic analysis for the Global Burden of Disease Study 2019. Lancet. 2021 Dec 19;396(10267):2006-2017. doi: 10.1016/S0140-6736(20)32340-0. Epub 2020 Dec 1. PMID 33275908
- [Background] van Hecke O, Torrance N, Smith BH. Chronic pain epidemiology and its clinical relevance. Br J Anaesth. 2013 Jul;111(1):13-8. doi: 10.1093/bja/aet123. PMID 23794640
- [Background] Mills S, Torrance N, Smith BH. Identification and Management of Chronic Pain in Primary Care: a Review. Curr Psychiatry Rep. 2016 Feb;18(2):22. doi: 10.1007/s11920-015-0659-9. PMID 26820898
- [Background] Hurwitz EL, Randhawa K, Yu H, Cote P, Haldeman S. The Global Spine Care Initiative: a summary of the global burden of low back and neck pain studies. Eur Spine J. 2018 Sep;27(Suppl 6):796-801. doi: 10.1007/s00586-017-5432-9. Epub 2018 Feb 26. PMID 29480409
- [Background] Chronic pain (primary and secondary) in over 16s: assessment of all chronic pain and management of chronic primary pain. London: National Institute for Health and Care Excellence (NICE); 2021 Apr 7. Available from http://www.ncbi.nlm.nih.gov/books/NBK569960/ PMID 33939353
- [Background] Korownyk CS, Montgomery L, Young J, Moore S, Singer AG, MacDougall P, Darling S, Ellis K, Myers J, Rochford C, Taillefer MC, Allan GM, Perry D, Moe SS, Ton J, Kolber MR, Kirkwood J, Thomas B, Garrison S, McCormack JP, Falk J, Dugre N, Sept L, Turgeon RD, Paige A, Potter J, Nickonchuk T, Train AD, Weresch J, Chan K, Lindblad AJ. PEER simplified chronic pain guideline: Management of chronic low back, osteoarthritic, and neuropathic pain in primary care. Can Fam Physician. 2022 Mar;68(3):179-190. doi: 10.46747/cfp.6803179. PMID 35292455
- [Background] Louw A, Diener I, Butler DS, Puentedura EJ. The effect of neuroscience education on pain, disability, anxiety, and stress in chronic musculoskeletal pain. Arch Phys Med Rehabil. 2011 Dec;92(12):2041-56. doi: 10.1016/j.apmr.2011.07.198. PMID 22133255
- [Background] Louw A, Zimney K, Puentedura EJ, Diener I. The efficacy of pain neuroscience education on musculoskeletal pain: A systematic review of the literature. Physiother Theory Pract. 2016 Jul;32(5):332-55. doi: 10.1080/09593985.2016.1194646. Epub 2016 Jun 28. PMID 27351541
- [Background] Stanton TR, Braithwaite FA, Butler D, Moseley GL, Hill C, Milte R, Ratcliffe J, Maher C, Tomkins-Lane C, Pulling BW, MacIntyre E, Esterman A, Stanford T, Lee H, Fraysse F, Metcalf B, Mouatt B, Bennell K. The EPIPHA-KNEE trial: Explaining Pain to target unhelpful pain beliefs to Increase PHysical Activity in KNEE osteoarthritis - a protocol for a multicentre, randomised controlled trial with clinical- and cost-effectiveness analysis. BMC Musculoskelet Disord. 2021 Aug 28;22(1):738. doi: 10.1186/s12891-021-04561-6. PMID 34454458
- [Background] Moseley GL, Butler DS. Fifteen Years of Explaining Pain: The Past, Present, and Future. J Pain. 2015 Sep;16(9):807-13. doi: 10.1016/j.jpain.2015.05.005. Epub 2015 Jun 5. PMID 26051220
- [Background] Van Oosterwijck J, Nijs J, Meeus M, Truijen S, Craps J, Van den Keybus N, Paul L. Pain neurophysiology education improves cognitions, pain thresholds, and movement performance in people with chronic whiplash: a pilot study. J Rehabil Res Dev. 2011;48(1):43-58. doi: 10.1682/jrrd.2009.12.0206. PMID 21328162
- [Background] Sillevis R, Trincado G, Shamus E. The immediate effect of a single session of pain neuroscience education on pain and the autonomic nervous system in subjects with persistent pain, a pilot study. PeerJ. 2021 May 31;9:e11543. doi: 10.7717/peerj.11543. eCollection 2021. PMID 34131526
- [Background] King R, Robinson V, Elliott-Button HL, Watson JA, Ryan CG, Martin DJ. Pain Reconceptualisation after Pain Neurophysiology Education in Adults with Chronic Low Back Pain: A Qualitative Study. Pain Res Manag. 2018 Sep 12;2018:3745651. doi: 10.1155/2018/3745651. eCollection 2018. PMID 30275918
- [Background] Galan-Martin MA, Montero-Cuadrado F, Lluch-Girbes E, Coca-Lopez MC, Mayo-Iscar A, Cuesta-Vargas A. Pain neuroscience education and physical exercise for patients with chronic spinal pain in primary healthcare: a randomised trial protocol. BMC Musculoskelet Disord. 2019 Nov 3;20(1):505. doi: 10.1186/s12891-019-2889-1. PMID 31679512
- [Background] Areso-Boveda PB, Mambrillas-Varela J, Garcia-Gomez B, Moscosio-Cuevas JI, Gonzalez-Lama J, Arnaiz-Rodriguez E, Del Barco MBA, Teodoro-Blanco PS. Effectiveness of a group intervention using pain neuroscience education and exercise in women with fibromyalgia: a pragmatic controlled study in primary care. BMC Musculoskelet Disord. 2022 Apr 4;23(1):323. doi: 10.1186/s12891-022-05284-y. PMID 35379222
- See also: Wilson et al are carrying out a study to detect the problems faced by physiotherapists practising freely in that country when applying interventions based on education in pain neuroscience. — https://www.noigroup.com/noijam/improving-pain-science-education-implementation-when-a-clinical-trial-isnt-enough/